CLINICAL TRIAL: NCT04503954
Title: Efficacy of Chronic Disease Self-management Program in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCHIRB-10904004
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Schizophrenia
Keywords: chronic disease self-management program
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management group (Experimental): Self-management group Chronic disease self-management program is conduct training skills, person how to live together with personal chronic disease to make life quality better.
  Interventions: Other: Chronic disease self-management program
- Control group (Placebo Comparator): Control group will continue general psychiatric intervention.
  Interventions: Other: General psychiatric intervention

INTERVENTIONS:
Other: Chronic disease self-management program — The chronic disease self-management program is based on the self-efficacy theory for improving health behavior, by the solve health problem skill, health life style, emotion management skill, improve intention of health condition in people with chronic disease.
  Arms: Self-management group
Other: General psychiatric intervention — General psychiatric intervention contains the activities in psychiatric center.
  Arms: Control group

SUMMARY:
This was a randomized controlled behavioral intervention trial to assess the efficacy of investigating program of chronic disease self-management program in people on schizophrenia patients conditions of depression, activities of daily living, social function, work, and quality of life.

DETAILED DESCRIPTION:
Subjects were randomized to intervention group and control group. The primary outcome included eight measures, Stanford Self-Management Questionnaire, the Beck Depression Inventory-II, the Activities of Daily Living Rating Scale III, the Instrumental Activities of Daily Living Scale, the Participation Measure-3 Domains, 4 Dimensions, the Work Behavior Inventory, and the Schizophrenia-Quality of Life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by DSM-5
* age > 20 years
* Stable mental symptoms
* Willing to sign the subject's consent

Exclusion Criteria:

* History of severe brain injury
* Substance abuse
* Diagnosis of intellectual developmental disorder
* Unable to follow instructions

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Stanford Self-Management Questionnaire | 6 week
  The Stanford Self-Management Questionnaire is for Chronic Disease Self-management Program. A higher score indicates better self-management. Changes of the Canadian Occupational Performance Measure will be assessed at the 0 week, 6 weeks.
Beck Depression Inventory-II, | 6 week
  Beck Depression Inventory-II assesses the person about depression. A higher score indicates more depression.
  Changes of Beck Depression Inventory-II will be assessed at the 0 week, 6 weeks.
Activities of Daily Living Rating Scale III, | 6 week
  Activities of Daily Living Rating Scale III assesses instrumental activities of daily living. A higher score indicates better activities of daily living. Changes of Activities of Daily Living Rating Scale III will be assessed at the 0 week, 6 weeks.
Instrumental Activities of Daily Living | 6 week
  Instrumental Activities of Daily Living assesses instrumental activities of daily living.
  A higher score indicates better instrumental activities of daily living. Changes of Instrumental Activities of Daily Living will be assessed at the 0 week, 6 weeks.
Participation Measure-3 Domains Domains, 4 Dimensions | 6 week
  Participation Measure-3 Domains, 4 Dimensions assesses social participation. A higher score indicates better social participation. Changes of Participation Measure-3 Domains, 4 Dimensions will be assessed at the 0 week, 6 weeks.
Work Behavior Inventory | 6 week
  Work Behavior Inventory assesses work behavior about chronic mental patients. A lower score indicates better work behavior. Changes of Work Behavior Inventory will be assessed at the 0 week, 6 weeks.
Schizophrenia-Quality of Life questionnaire | 6 week
  Schizophrenia-Quality of Life questionnaire assesses schizophrenia quality of life. A higher score indicates better quality of life. Changes of Schizophrenia-Quality of Life questionnaire will be assessed at the 0 week, 6 weeks.
Mini Mental State Examination-2nd edition | 6 week
  Mini Mental State Examination general cognitive function. A higher score indicates better general cognitive function.
  Changes of Mini Mental State Examination will be assessed at the 0 week, 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: En-Chi Chiu, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Wanhua Dist, Taiwan